CLINICAL TRIAL: NCT04416139
Title: Mesenchymal Stem Cells for the Treatment of Severe Acute Respiratory Distress Syndrome Due to COVID-19. Pilot Study
Brief Title: Mesenchymal Stem Cell for Acute Respiratory Distress Syndrome Due for COVID-19
Acronym: COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Martín Iglesias, Plastic surgeon, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI-3354-20-21-1
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Covid 19
Keywords: Mesenchymal Stem Cell
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Mesenchymal Stem Cell from umbilical cord allogenic from de bank laboratory, will be applied IV to 5 patients con pneumonia bilateral due to COVID 19, complicated with acute respiratory distress syndrome. The clinical, biochemical, inflammatory and immune changes will be described and compare against historical cases treated in the Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Active Comparator): Five patients, of any sex and age, with bilateral COVID-19 pneumonia, severe SIRA with PaO2 / FiO2 less than 150, lymphopenia less than 800 total lymphocytes, CT with bilateral pneumonia, SOFA less than 11 and that has not improved in relation to the following parameters: a) persistent PaO2 / FiO2 less than 150; b) persistent fever, c) increase in D-dimer of at least 50% of the baseline and / or ferritin greater than 1000, after 48 h of hospital stay receiving the standard management measures used at that time in the Care Center, will be included in the study. This treatment will be administered after discussing it with the relatives that it is a procedure considered as rescue and will be carried out with informed consent.
  Interventions: Biological: Infusion IV of Mesenchymal Stem cells
- Control Group (No Intervention): The results obtained in the treated group will be compared against the historical controls treated in INCMNSZ, evaluating the same variables.

INTERVENTIONS:
Biological: Infusion IV of Mesenchymal Stem cells — Mesenchymal Stem cells from bank will be applied IV, at dose 1 million xKg in a single dose
  Arms: Treated group

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is the main cause of death from COVID-19. One of the main mechanisms for ARDS is the violent storm of cytokines and chemokines, which cause uncontrolled fatal systemic inflammation by the immune system on the body, with additional multiple organ failure. Mortality in cases of severe ARDS caused by COVID 19 varies significantly between 50 and 90%, basically depending on the age of the patient and the presence of comorbidities.

The plasticity of Mesenchymal Stem Cells (MSC) regulates inflammation and immunity. MSC can promote and inhibit an immune response, depending on the dynamics of inflammation and depending on the activation force of the immune system, the types of inflammatory cytokines present, and the effects of immunosuppressants. Essentially, the state of inflammation determines the immunoregulatory fate of MSC. Thus, IV application of AMSCa has been shown to control the inflammatory response in various diseases, such as the graft-versus-host reaction and the ARDS caused by H5NI.

The objective of this study is to describe the clinical changes secondary to IV administration of MSC allogenic, in patients with bilateral COVID-19 pneumonia complicated by severe ARDS, with the evaluation of the PaO2 / FiO2 ratio, heart and respiratory rates, and the fever curve.

Five patients, of either sex, over 18 years of age, with bilateral pneumonia caused by COVID-19 and severe SIRA that has not improved with the standard management measures used at that time in the care center, will be included in the study. This treatment will be administered after discussing it with the relatives that it is a procedure considered as rescue and will be carried out with informed consent. 1x10(6) xKg will be applied IV.

The follow-up of the patient will be for three weeks. PaO2 / FiO2 data, fever, inflammatory markers and immunity will be evaluated. The results will be compared with the historical controls attended at INCMNSZ.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is the main cause of death from COVID-19. One of the main mechanisms for ARDS is the storm of cytokines and chemokines, which cause uncontrolled fatal systemic inflammation. The SARS-CoV-2 virus infects cells that express the angiotensin II converting enzyme receptor (ACE2). This receptor is widely distributed on the surface of type II alveolar cells (AT2) and on the capillary endothelium. This is why the cytokine storm will trigger a violent attack by the immune system on the body, cause ARDS and multiple organ failure, and can ultimately lead to death. Mortality in cases of severe SIRA caused by COVID 19 varies significantly between 50 and 90%, basically depending on the age of the patient and the presence of comorbidities.

The plasticity of Mesenchymal Stem Cell (MSC) regulates inflammation and immunity. MSC can promote and inhibit an immune response, depending on the dynamics of inflammation and depending on the activation force of the immune system, the types of inflammatory cytokines present, and the effects of immunosuppressants. Essentially, the state of inflammation determines the immunoregulatory fate of MSC. Thus, IV application of MSC has been shown to control the inflammatory response in various diseases, such as the graft-versus-host reaction and the ARDS caused by H5NI.

MSC are negative for ACE2, therefore they have been used to decrease the cytokine storm present in COVID-19.

Two recent studies in China have used human allogeneic MSC to treat COVID-19 pneumonia. Both studies reveal a marked reversal of symptoms, even in critically serious cases. Lung function improved two days after MSC application and 10 days later they were discharged. Lymphocytes increased, PCR decreased, and cytokine-producing immune cells disappeared within 3 to 6 days. Regulatory immune cells increased. TNF alpha factor decreased and IL10 increased.

Taking into account the previous concepts together with the current global pandemic, and the high mortality existing among patients with bilateral pneumonia caused by COVID-19 and severe ARDS, the investigators propose intravenous infusion of mesenchymal stem cells from bank laboratory, with the purpose partially proven to decrease the systemic inflammatory process, offering it as a salvage treatment.

Five patients, of either sex, over 18 years of age, with bilateral pneumonia caused by COVID-19 and severe ARDS that has not improved in relation to the following parameters: a) Persistent PaO2 / FiO2 less than 150, b) persistent fever, c ) D-dimer increase of at least 50% of baseline and / or ferritin greater than 1000, after 48 h of hospital stay receiving the standard management measures used at that time in the care center, will be included in the study. Covid pneumonia should be confirmed by chest CT and RNA detection by positive SARS-Cov2 PCR. This treatment will be administered after discussing it with the relatives that it is a procedure considered as rescue and will be carried out with informed consent.

Their follow-up will be daily while they are hospitalized in the Intensive Care Unit and / or hospitalized, until their discharge from the hospital or until the third week after surgery. If the patient has already been discharged from the hospital, his last evaluation will be in the third week.

The main objective of this protocol is: To describe the clinical changes secondary to IV administration of MSC, in patients with bilateral COVID-19 pneumonia complicated by severe ARDS, with the evaluation of the PaO2 / FiO2 ratio, heart rate and respiratory rate, as well as of the fever curve daily.

The secondary objectives are:

a) To assess the effect of the proposed treatment on the general biochemical indicators (Leukocytes, absolute lymphocytes, absolute neutrophils, absolute monocytes, absolute eosinophils, absolute basophils, erythrocytes, hemoglobin, platelets, total bilirubin, albumin, amino-aspartate transferase, fibrinogen, procalcitonin, glomerular filtration, myoglobin, troponin, ferritin and D-dimer. Daily.

b. To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of cytokines, and C-reactive protein, TNFa, IL10, IL1, IL6, IL17, VEGF in plasma. These variables will be evaluated before treatment, upon discharge from the ICU, and / or from the Hospital.

c. Assess the radiological evolution of the proposed treatment through simple chest CT. These variables will be evaluated before treatment, upon discharge from the ICU, and / or from the Hospital.

d. Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: regulatory T cells (CXCR3-), dendritic cells (DC, CXCR3-), CXCR3 + CD4 + T, CXCR3 + CD + T, and CXCRT3 + NK. These variables will be evaluated before treatment, upon discharge from the ICU, and / or from the Hospital.

e) Assess the safety of the proposed treatment (allergic reactions and / or infection) F. To assess the negativization of the RNA detection test by SARS-Cov2 PCR. These variables will be evaluated before treatment, upon discharge from the ICU, and / or from the Hospital.

The inclusion criteria are:

1. Comply with the informed consent procedure and sign the informed consent form.
2. Over 18 years
3. Of any gender
4. With SARS-Cov2 PCR RNA detection test, positive
5. With bilateral pneumonia caused by COVID-19
6. Severe ARDS with PaO2 / FiO2 less than 150
7. That it has not improved in relation to: a) Persistent PaO2 / FiO2 less than 150, b) persistent fever, c) increase in D-dimer at least 50% of the baseline and / or ferritin greater than 1000, after 48 hrs hospital stay receiving the standard management measures used at that time in the care center.
8. Lymphopenia less than 800 total lymphocytes
9. Increased D-dimer (> 1200 mg / dl)
10. CT compatible with bilateral pneumonia
11. SOFA under 11 With knowledge of the patient and / or their responsible relatives that it is a rescue treatment, in an experimental phase.

The bank mesenchymal cells will be donated by the CBCells Bio Technology Laboratory, at no cost to the patient or INCMNSZ.

1x106 x Kg of weight, diluted in 100 ml of saline, will be infused intravenously, to pass in 40 minutes. It will be monitored with monitors, Pao2 / Fio2, FC, FR, ECG. Additionally, fever and muscle contractures will be monitored, which will be recorded every hour for 24 hours and every 24 hours thereafter, up to three weeks after the application of MSC. The patient should continue with their indicated medical treatments, such as antibiotics and specific treatments in case of comorbidities.

The results will be compared with the historical controls attended at INCMNSZ Thus, the results obtained will give information to calculate the sample size in subsequent studies in which the usefulness of the procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral pneumonia due to COVID-19
* With SARS-Cov2 PCR RNA detection test, positive
* Severe ARDS
* PaO2/FiO2 <150
* Leukocytes < 800
* Chest TAC with pneumonia bilateral
* persistant fever
* increase 50% D-Dimer, respect to basal value
* Ferritin > 1000
* SOFA < 11
* Medical treatment during 48 hr according to de Institutional Medical center
* With knowledge of the patient and / or his relatives responsible that it is a rescue treatment, in experimental phase.

Exclusion Criteria:

* Pneumonia or ARDS caused by COVID-19, mild and moderate.
* More than three organic failures
* Expectations of survival less than 48 hr in the opinion of the treating service
* Pneumonia or SIRA not caused by COVID-19
* Advance will of the patient to refuse rescue or experimental treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Functional Respiratory changes: PaO2 / FiO2 ratio | Three weeks
  To describe the clinical changes secondary to IV administration of AMSCa, in patients with bilateral COVID-19 pneumonia complicated by severe SIRA, with the evaluation of the PaO2 / FiO2 ratio.
Clinical cardiac changes: Heart rate per minute | Three weeks
  To describe the clinical changes secondary to IV administration of AMSCa, in patients with bilateral COVID-19 pneumonia complicated by severe SIRA, with the evaluation of the heart rate per minute.
Clinical Respiratory Changes: Respiratory rate per minute | Three weeks
  To describe the clinical changes secondary to IV administration of AMSCa, in patients with bilateral COVID-19 pneumonia complicated by severe SIRA, with the evaluation of the respiratory rate per minute.
Changes in body temperature | Three weeks
  To describe the clinical changes secondary to IV administration of AMSCa, in patients with bilateral COVID-19 pneumonia complicated by severe SIRA, with the evaluation of the fever curve in degrees centigrade.

SECONDARY OUTCOMES:
General biochemical changes in Leukocytes | Three weeks
  To assess the effect of the proposed treatment on the total Leukocytes
General biochemical changes on lymphocytes | Three weeks
  To assess the effect of the proposed treatment on absolute lymphocytes
General biochemical changes on platelets | Three weeks
  To assess the effect of the proposed treatment on total platelets
General biochemical changes on fibrinogen | Three weeks
  To assess the effect of the proposed treatment on serum fibrinogen
General biochemical changes on pocalcitonin | Three weeks
  To assess the effect of the proposed treatment on procalcitonin
General biochemical changes on ferritin | Three weeks
  To assess the effect of the proposed treatment on ferritin
General biochemical changes on D-dimer | Three weeks
  To assess the effect of the proposed treatment on D-dimer
Changes on inflammatory C-reactive protein | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of C-reactive protein
Cahnges on Inflammatory cytokine TNFa | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of TNFa in plasma.
Changes on Inflammatory cytokine IL10 | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of IL10 in plasma.
Changes on Inflammatory cytokine IL1 | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of IL1 in plasma.
Changes on Inflammatory cytokine IL6 | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of IL6 in plasma.
Changes on Inflammatory cytokine IL 17 | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of IL17 in plasma
Changes on VEGF | Three weeks
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of VEGF in plasma
Radiological Changes | Three weeks
  Assess the radiological evolution of the proposed treatment through simple chest CT
Immunological changes on T cell | Three weeks
  Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: regulatory T cells
Immunological changes on Dendritic cells | Three weeks
  Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: dendritic cells
Immunological changes on CD4+ T | Three weeks
  Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: CD4 + T
Immunological changes on CD8+ T | Three weeks
  Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: CD8 + T
Immunological changes on NK cell | Three weeks
  Evaluate immune system improvement with mass cytometry to analyze patients' immune cells: NK cells
Adverse events | Three weeks
  Evaluate the safety of the proposed treatment (allergic reactions and / or infection)
RNA detection by SARS-Cov2 PCR | Three weeks
  To assess the negativization of the SARS-Cov2 PCR RNA detection test

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No